CLINICAL TRIAL: NCT01774565
Title: A Randomised Study to Assess the Efficacy and Safety of Automated Closed-loop Glucose Control in Insulin Treated Type 2 Diabetes (Phase 1), Inpatient Hyperglycaemia Requiring Subcutaneous Insulin Therapy (Phase 2 and Phase 3) and to Evaluate Use of Closed-loop Applying Faster Insulin Aspart Versus Standard Insulin Aspart (Phase 4)
Brief Title: Closed-loop Insulin Delivery in the General Ward
Acronym: ANGIE02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Hood Thabit, Clinical Investigator, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANGIE02; A092763 (Other: R&D Office, Cambridge University Hospitals NHS Foundation Trust)
Record Dates: First submitted 2013-01-18; First posted 2013-01-24 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Insulin; Closed-Loop; Real-time CGM; Subcutaneous insulin pump; Hospital
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomised parallel (phase 1-3) and randomised crossover (phase 4)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fully Automated Closed-Loop Insulin Delivery (phase 1-4) (Experimental): The control algorithm will automatically direct between meals and meal-related subcutaneous insulin delivery utilizing real-time continuous glucose monitoring (RT-CGM) data. The subcutaneous insulin pump will deliver insulin Aspart or similar. In phase 1, a once daily basal insulin analogue will also be given subcutaneously at 20% the patient's usual total daily dose. In phase 3 and 4 faster-acting insulin aspart (Fiasp) is applied.
  Interventions: Device: Fully Automated Closed-Loop Insulin Delivery
- Usual care/ fully-automated closed-loop using Iasp (Active Comparator): Phase 1-3: During usual care (conventional therapy), subject's s.c. insulin dose and regimen on admission will be adjusted as necessary by the clinical team according to local centres' usual clinical practice. Subjects will have masked CGM sensors inserted during the study (CGM readings will be masked throughout the study).
  Phase 4: subjects will receive fully-automated insulin delivery using standard insulin aspart (Iasp)
  Interventions: Device: Conventional insulin therapy

INTERVENTIONS:
Device: Fully Automated Closed-Loop Insulin Delivery
  Arms: Fully Automated Closed-Loop Insulin Delivery (phase 1-4)
Device: Conventional insulin therapy
  Arms: Usual care/ fully-automated closed-loop using Iasp

SUMMARY:
The study assesses the efficacy and safety of closed-loop glucose control in patients with insulin-treated type 2 diabetes.

Phase 1 The study objective is to compare conventional insulin therapy with closed-loop glucose control combined with once daily basal insulin injection over 72 hours in hospitalised insulin treated T2D subjects.

Phase 2 The study objective is to compare conventional insulin therapy with closed-loop glucose control up to maximum 15 days in hospitalised insulin treated T2D subjects.

Phase 3 The study objective is to compare conventional insulin therapy with closed-loop glucose control applying faster insulin aspart up to maximum 15 days in insulin-treated inpatients receiving parenteral and/or enteral nutrition.

Phase 4 The study objective is to compare automated closed-loop control using faster acting insulin aspart with closed-loop control using standard insulin aspart.

DETAILED DESCRIPTION:
Hyperglycaemia in hospitalized patients is becoming a common clinical problem due to the increasing prevalence of diabetes mellitus . Hyperglycaemia in this cohort can also occur in patients with previously undiagnosed diabetes, or during acute illness in those with previously normal glucose tolerance. As a result, the prevalence of acute or stress hyperglycaemia in hospitalised patients has been widely reported. A growing body of evidence currently suggest that the degree of hyperglycaemia upon admission and the duration of hyperglycaemia during their illness are associated with adverse outcomes.In-patient hyperglycaemia is now widely recognised as a poor prognostic marker in terms of morbidity and mortality, increased length of stay and cost to the healthcare system.

The current management of in-patient hyperglycaemia in non-critical care is still far from ideal, and vary widely between different centres. The discordance between clinical evidence and practice is due to a number of factors which could potentially undermine patient care and safety. Of these, hypoglycaemia remains one the biggest barriers to managing in-patient hyperglycaemia. There is therefore a need to develop and validate a more effective and safer system to manage in-patient hyperglycaemia.

A closed-loop insulin infusion system has previously been tested and reported to be feasible and safe in intensive care patients. Its utilisation in non-critical patients in the general medical and surgical wards currently remains unproven. Its use in this cohort however could potentially be of significant practical and clinical value, especially in a busy ward environment. The Model Predictive Control (MPC) algorithm developed by our group at the University of Cambridge utilises fundamental glucoregulatory processes and predicts future glucose excursion resulting from projected insulin infusion rates. The algorithm can also account for the patient's meal intake and the duration of action of the short acting insulin used. This has the distinct advantage over the "reactive" approach of sliding scale insulin protocols, which treats hyperglycaemia after it has already occurred.

The MPC algorithm has been studied in intensive care and cardiac surgery patients, and results from these studies to date have been encouraging. It is shown to be associated with a significantly higher percentage of time within the blood glucose target range, without increasing the risk of severe hypoglycaemia. The expectant role of a closed-loop system using the MPC algorithm in non-critical care patients would therefore be to provide clinicians with an effective and safe method to manage hyperglycaemia in hospital.

In early 2017, faster-acting insulin aspart (Fiasp, Novo Nordisk, Copenhagen, Denmark) received marketing authorisation from the European Commission. Due to the more favourable pharmacokinetic profile, Fiasp has the potential to further improve safety and efficacy of fully automated closed-loop glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Type 2 Diabetes for at least 1 year as defined by WHO (phase 1 and 4)
* Inpatient hyperglycaemia requiring subcutaneous insulin therapy (phase 2 and 3)
* Treatment with subcutaneous insulin alone or in combination with oral glucose-lowering medication(s) (phase 4: basal bolus insulin regime for at least 3 months)
* Receiving parenteral and/or enteral nutrition (phase 3)
* HbA1c<11.0% (phase 4)

Exclusion Criteria:

* Autoimmune type 1 diabetes
* Known or suspected allergy against insulin
* Known proliferative retinopathy
* Current or planned pregnancy or breast feeding
* Unstable or end-stage cardiac and renal disease (phase 1 only)
* Planned surgery during study period (phase 1 only)
* Current in-patient in intensive care unit
* Any physical or psychological disease or medication(s) likely to interfere with the conduct of the study and interpretation of the study results, as judged by the study clinician
* Likely discharge earlier than 72 hours (phase 1 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Time spent in target glucose range (5.6-10.0mmol/l) | Phase 1 (Pilot study) = 72-hours, Phase 2 (Follow-up study) = Up to 15 days
  Primary outcome will be measured using continuous subcutaneous glucose monitoring (CGM) data (Phase 1-3) and plasma (Phase 4).

SECONDARY OUTCOMES:
Proportion of time with glucose levels below 5.6 mmol/l and above 10.0 mmol/l as recorded by CGM | Phase 1 (Pilot study) = 72-hours, Phase 2 and Phase 3 (Follow-up study)= Up to 15 days, Phase 4=between 07:00 and 17:00
  CGM (Phase 1-4) and plasma glucose (Phase4)
Average glucose levels, as recorded by CGM | Phase 1 (Pilot study) = 72-hours, Phase 2 and Phase 3 (Follow-up study)= Up to 15 days, Phase 4=between 07:00 and 17:00
  CGM (Phase 1-4) and plasma glucose (Phase4)
Proportion of time with glucose levels below 3.9 mmol/l as recorded by CGM | Phase 1 (Pilot study) = 72-hours, Phase 2 and Phase 3 (Follow-up study)= Up to 15 days, Phase 4=between 07:00 and 17:00
  CGM (Phase 1-4) and plasma glucose (Phase4)
Proportion of time with glucose levels below 3.0 mmol/l as recorded by CGM | Phase 2 and Phase 3 (Follow-up study)= Up to 15 days, Phase 4= over 10 hours
  CGM (Phase 1-4) and plasma glucose (Phase4)
Proportion of time with glucose levels below 2.8 mmol/l as recorded by CGM | Phase 2 and Phase 3 (Follow-up study)= Up to 15 days, Phase 4= over 10 hours
  CGM (Phase 1-4) and plasma glucose (Phase4)
Area under the curve of sensor glucose levels below 3.5 mmol/l as recorded by CGM | Phase 1 (Pilot study) = 72-hours, Phase 2-3 (Follow-up study) = Up to 15 days, Phase 4= over 10 hours
  CGM (Phase 1-4) and plasma glucose (Phase4)
Area under the curve of sensor glucose levels below 3.0 mmol/l as recorded by CGM | Phase 2-3 (Follow-up study) = Up to 15 days, Phase 4= over 10 hours
  CGM (Phase 1-4) and plasma glucose (Phase4)
Standard deviation and coefficient of variation of glucose levels, as recorded by CGM | Phase 1 (Pilot study) = 72-hours, Phase 2-3 (Follow-up study) = Up to 15 days, Phase 4= over 10 hours
  CGM (Phase 1-4) and plasma glucose (Phase4)
Proportion of time with glucose levels in significant hyperglycaemic range (>20mmol/l) as recorded by CGM | Phase 2-3 (Follow-up study) = Up to 15 days, Phase 4= over 10 hours
  CGM (Phase 1-4) and plasma glucose (Phase4)
Total daily insulin dose | Phase 2-3 (Follow-up study) = Up to 15 days, Phase 4= over 10 hours
Between 24 hour period variability | Phase 2-3 (Follow-up study) = Up to 15 days, Phase 4= over 10 hours
  Coefficient of variation of CGM glucose between 24 hour periods (08:00 to 08:00) (Phase 1-3)
Number of capillary glucose confirmed hypoglycaemic events <3.5mmol/l | Phase 2-3 (Follow-up study) = Up to 15 days, Phase 4= over 10 hours
  Capillary glucose measurements will be performed using hospital point of care devices
Pre-breakfast, pre-lunch, pre-dinner, and evening capillary glucose values | Phase 2-3 (Follow-up study) = Up to 15 days
  Capillary glucose measurements will be performed using hospital point of care devices (Phase 1-3)

OTHER OUTCOMES:
Overnight period: Proportion of time with Glucose levels in target range (5.6-10.0mmol/l) as recorded by CGM | Phase 2-3 (Follow-up study) = Up to 15 days
  Between 24:00 and 08:00
Overnight period: Average glucose levels, as recorded by CGM | Phase 2-3 (Follow-up study) = Up to 15 days
  Between 24:00 and 08:00
Overnight period: Standard deviation and coefficient of variation of glucose levels, as recorded by CGM | Phase 2-3 (Follow-up study) = Up to 15 days
  Between 24:00 and 08:00
Overnight period: Area under the curve of sensor glucose levels below 3.5 mmol/l as recorded by CGM | Phase 2-3 (Follow-up study) = Up to 15 days
  Between 24:00 and 08:00
Between night variability | Phase 2-3 (Follow-up study) = Up to 15 days
  Coefficient of variation of CGM glucose between nights (24:00 and 08:00 ) (Phase 1-3)
Total insulin dose overnight | Phase 2-3 (Follow-up study) = Up to 15 days
  Closed-loop only (24:00 and 08:00 ) (Phase 1-3)
Day period: Proportion of time with glucose levels in target range (5.6-10.0mmol/l) as recorded by CGM | Phase 2-3 (Follow-up study) = Up to 15 day
  Between 08:00 and 24:00 (Phase 1-3)
Day period: Average glucose levels, as recorded by CGM | Phase 2-3 (Follow-up study) = Up to 15 day
  Between 08:00 and 24:00 (Phase 1-3)
Day period: Standard deviation and coefficient of variation of glucose levels, as recorded by CGM | Phase 2-3 (Follow-up study) = Up to 15 day
  Between 08:00 and 24:00 (Phase 1-3)
Day period: Area under the curve of sensor glucose levels below 3.5 mmol/l as recorded by CGM | Phase 2-3 (Follow-up study) = Up to 15 day
  Between 08:00 and 24:00 (Phase 1-3)
Between day variability | Phase 2-3 (Follow-up study) = Up to 15 day
  Coefficient of variation of CGM glucose between days (08:00 and 24:00 ) (Phase 1-3)
Total insulin dose during the day | Phase 2-3 (Follow-up study) = Up to 15 days
  Closed-loop only (08:00 and 24:00 ) (Phase 1-3)
Safety: Number of subjects and number of occurences of severe hypoglycaemic events (capillary glucose <2.2mmol/l) | Phase 2-3 (Follow-up study) = Up to 15 days, Phase 4 = up to 4 weeks
Safety: Significant hyperglycaemic events (capillary glucose >20mmol/l) with or without ketonaemia (B-OHB >0.6mmol/l) | Phase 2 (Follow-up study) = Up to 15 days, Phase 4 = up to 4 weeks
Safety: Number of other (serious) adverse events (including adverse device effects) and device deficiencies | Phase 2 (Follow-up study) = Up to 15 days, Phase 4 = up to 4 weeks
2-hour postprandial incremental plasma glucose (Phase 4 only) | 120min after meal intake
  CGM and plasma glucose
Peak glucose (Phase 4 only) | over 10 hours
  CGM and plasma glucose
Mean insulin concentration (Phase 4 only) | over 10 hours
  Plasma insulin concentration
Time to maximal insulin concentration (Phase 4 only) | over 10 hours
  Time (min) to maximal plasma insulin concentration
Maximal insulin concentration (Phase 4 only) | over 10 hours
  Maximal plasma insulin concentration
Total and endogenous insulin exposure within 1 hour postprandial period (Phase 4 only) | over 10 hours
  Total and endogenous plasma insulin exposure within 1 hour post-meal (iAUC)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, MSc, BSc, Principal Investigator — University of Cambridge
Locations (2):
- Inselspital, Bern University Hospital, University of Bern, Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Bern, Switzerland
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

REFERENCES:
- [Derived] Bally L, Gubler P, Thabit H, Hartnell S, Ruan Y, Wilinska ME, Evans ML, Semmo M, Vogt B, Coll AP, Stettler C, Hovorka R. Fully closed-loop insulin delivery improves glucose control of inpatients with type 2 diabetes receiving hemodialysis. Kidney Int. 2019 Sep;96(3):593-596. doi: 10.1016/j.kint.2019.03.006. Epub 2019 Mar 20. PMID 31133457
- [Derived] Boughton CK, Bally L, Martignoni F, Hartnell S, Herzig D, Vogt A, Wertli MM, Wilinska ME, Evans ML, Coll AP, Stettler C, Hovorka R. Fully closed-loop insulin delivery in inpatients receiving nutritional support: a two-centre, open-label, randomised controlled trial. Lancet Diabetes Endocrinol. 2019 May;7(5):368-377. doi: 10.1016/S2213-8587(19)30061-0. Epub 2019 Mar 29. PMID 30935872
- [Derived] Bally L, Thabit H, Hartnell S, Andereggen E, Ruan Y, Wilinska ME, Evans ML, Wertli MM, Coll AP, Stettler C, Hovorka R. Closed-Loop Insulin Delivery for Glycemic Control in Noncritical Care. N Engl J Med. 2018 Aug 9;379(6):547-556. doi: 10.1056/NEJMoa1805233. Epub 2018 Jun 25. PMID 29940126
- [Derived] Thabit H, Hartnell S, Allen JM, Lake A, Wilinska ME, Ruan Y, Evans ML, Coll AP, Hovorka R. Closed-loop insulin delivery in inpatients with type 2 diabetes: a randomised, parallel-group trial. Lancet Diabetes Endocrinol. 2017 Feb;5(2):117-124. doi: 10.1016/S2213-8587(16)30280-7. Epub 2016 Nov 9. PMID 27836235